CLINICAL TRIAL: NCT04085081
Title: Feasibility of a Perioperative Physical Activity Intervention for Older Adults With Lung Cancer and Their Family Caregivers
Brief Title: Physical Activity Intervention Before and After Surgery in Older Adults With Lung Cancer and Their Family Caregivers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issue
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19252; NCI-2019-05582 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19252 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Caregiver; Lobectomy Patient; Lung Carcinoid Tumor; Lung Non-Small Cell Carcinoma
Keywords: Lung cancer; geriatric oncology; physical activity; family caregivers; functional status
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Motor Activity | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (coaching call, motivational messages) (Experimental): Patients and family caregivers complete comprehensive geriatric and functional assessments before surgery. This information is used to develop a personalized walking program plus simple lower extremity strength exercises. The intervention is administered by trained coaches with physical and occupational therapy background. The sessions are delivered by telephone before surgery (30-60 minutes), and on days 2, 7, 14, and 21 after hospital discharge (20-50 minutes). Participants will also receive brief motivational text or email messages (4 times per week between telephone sessions) to provide support, promote physical activity behavior change, and to sustain participant engagement.
  Interventions: Other: E-mail; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention; Other: Text Message

INTERVENTIONS:
Other: E-mail — Receive brief motivational text or email messages
  Other Names: Electronic Mail; Email
Behavioral: Exercise Intervention — Receive personalized walking program plus strength exercises
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive intervention coaching sessions via telephone
Other: Text Message — Receive brief motivational text or email messages
  Other Names: SMS Text; SMS Text Message; Text

SUMMARY:
This trial studies whether a telephone-based physical activity intervention before and after lung cancer surgery can be provided to older patients and their caregivers. The trial also aims to understand whether patients and family caregivers will be satisfied with the intervention. Participating in physical activity such as walking before and after lung cancer surgery may improve functional status and recovery in older patients and their family caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Administer and determine the feasibility of the perioperative physical activity intervention.

SECONDARY OBJECTIVES:

I. To describe patient and family caregiver outcome patterns and trajectory pre- and post-intervention.

II. Using qualitative methods, evaluate the acceptability of the intervention through brief, semi-structured interviews with patients and family caregivers.

OUTLINE:

Patients and family caregivers complete comprehensive geriatric and functional assessments before surgery. This information is used to develop a personalized walking program plus simple lower extremity strength exercises. The intervention is administered by trained coaches with physical and occupational therapy background. The sessions are delivered by telephone before surgery (30-60 minutes), and on days 2, 7, 14, and 21 after hospital discharge (20-50 minutes). Participants will also receive brief motivational text or email messages (4 times per week between telephone sessions) to provide support, promote physical activity behavior change, and to sustain participant engagement.

Patients and family caregivers are followed up to day 30 after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Must have histologically confirmed non-small cell lung cancer (NSCLC) or carcinoid tumor of the lung, and registration must occur after the first histologic diagnosis
* PATIENTS: Must be registered at least 15 days before their scheduled surgery
* PATIENTS: Must be scheduled for a lobectomy (open or minimally invasive)
* PATIENTS: Must have access to a smartphone or telephone for study intervention sessions and study text messages
* PATIENTS: Age >= 70 years
* PATIENTS: Must be willing to wear a wristband pedometer for the duration of the study period, except on day of surgery
* PATIENTS: Must be willing to answer telephone calls from the City of Hope Call Center
* PATIENTS: Must have an identified family member or friend who is enrolled in the study
* PATIENTS: Able to read and comprehend English. Study materials and telephone calls are only available in English
* FAMILY CAREGIVERS: Family member or friend identified by the patient and will be caring for the patient before and after surgery
* FAMILY CAREGIVERS: Age >= 18 years
* FAMILY CAREGIVERS: Must have access to a smartphone or telephone for study intervention sessions and study text messages
* FAMILY CAREGIVERS: Must be willing to wear a wristband pedometer for the duration of the study period
* FAMILY CAREGIVERS: Must be willing to answer telephone calls from the City of Hope Call Center
* FAMILY CAREGIVERS: Must have a care recipient (patient) who is enrolled in the study
* FAMILY CAREGIVERS: Able to read and comprehend English. Study materials and telephone calls are only available in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment of >= 70% of eligible participants | Up to 30 days post-hospital discharge
  Will be evaluated based on data obtained throughout the study. Descriptive statistics will be assessed using means, standard deviations, and ranges for continuous variables, and frequencies and percentages for categorical variables.
>= 70% of enrolled participants who answer the telephone calls from City of Hope interventionists | Up to 30 days post-hospital discharge
  Will be evaluated based on data obtained throughout the study. Descriptive statistics will be assessed using means, standard deviations, and ranges for continuous variables, and frequencies and percentages for categorical variables.
Adherence/engagement | Up to 30 days post-hospital discharge
  Will be determined by >= 70% of enrolled participants who complete at least 2 intervention sessions. Descriptive statistics will be assessed using means, standard deviations, and ranges for continuous variables, and frequencies and percentages for categorical variables.

SECONDARY OUTCOMES:
Intervention acceptability as reported by participants | Up to 30 days post-hospital discharge
  Acceptability will be assessed through qualitative data analysis of exit interviews using content analysis approach.

OTHER OUTCOMES:
Patient and family caregiver outcome patterns and trajectories before and after the intervention | Baseline up to 30 days post-hospital discharge
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to explore patterns and trajectories over time.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center